CLINICAL TRIAL: NCT05177874
Title: Multicentric, Prospective, Controlled, Randomised Clinical Study of the Device Traumacel FAM Trium in the Post-market Surveillance Phase
Brief Title: Traumacel FAM Trium in the Post-market Surveillance Phase
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bioster, a.s. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PMCF-29-11-19
Record Dates: First submitted 2021-12-01; First posted 2022-01-05 (Actual); Last update posted 2022-01-05 (Actual); Status verified 2021-12

CONDITIONS: Bleeding; Surgical Wound
Keywords: Oxidized cellulose; Haemostatic agent
MeSH Terms: conditions — Hemorrhage; Surgical Wound

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traumacel FAM Trium (Experimental): Randomized application haemostatic agent Traumacel FAM Trium in the bleeding site.
  Interventions: Device: Traumacel FAM Trium
- Surgicel Fibrillar (Active Comparator): Randomized application of haemostatic agent Surgicel Fibrillar in the bleeding site.
  Interventions: Device: Surgicel Fibrillar

INTERVENTIONS:
Device: Traumacel FAM Trium — Absorbable Hemostat (oxidized non-regenerated cellulose)
  Other Names: Traumastem FAM Trium; EMOXICEL FAM Trium; Traumastem Fibrillar; Celstat Fibrillar
  Arms: Traumacel FAM Trium
Device: Surgicel Fibrillar — Absorbable Hemostat (oxidized regenerated cellulose)
  Arms: Surgicel Fibrillar

SUMMARY:
The investigational medical device Traumacel FAM Trium is a sterile plant polysaccharide haemostatic agent based on the oxidized cellulose in the form of multilayer nonwoven fabric. It is used as an adjunct to stop capillary, venous, or small arterial bleeding, and also to prevent early postoperative bleeding. It can be used in all areas of stopping diffuse bleeding from resection surfaces such as parenchymatous organs, muscles or defined body cavities. The wide scope of application allows the use for classical, robotic surgery and endoscopic treatments (e.g. laparoscopic).

The main objective of the study is to compare the efficacy and safety of Traumacel FAM Trium and regenerated oxidized cellulose based fibrous haemostat when used in accordance with their intended purpose. The partial objectives are: identification of any previously unknown side-effects and monitoring of known side-effects; identification and analysis of potentially newly emerging risks; confirmation of the acceptability of the benefit-risk ratio; identification of any systematic misuse of the device or off-label use of the device in order to verify the correctness of its intended purpose.

ELIGIBILITY:
Inclusion Criteria:

* Minimum age of 18.
* Surgical intervention.
* Negative pregnancy test of women in fertile age.
* Diffuse soft tissue, vascular or parenchymal haemorrhage after conventional surgical haemostatic methods have not worked or are impractical (e.g. ligation, suture, compression, cauterisation).
* Informed consent

Exclusion Criteria:

* Hypersensitivity or a known reaction to oxidized cellulose.
* Age under 18
* A severe clinical condition of the patient (e.g. associated illness, mental disorder) which, according to the investigator, could adversely affect patient safety and/or compliance with the procedures used in the study.
* The patient has participated in another clinical study involving a haemostatic product within 30 days prior to enrolment, or another such clinical study is planned during the subject's participation in the study.
* Pregnancy or lactation.
* If during the procedure itself, there was no need to use the test agent
* Application of any other topical haemostatic product prior to application of the test agent to the same site.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2020-05-18 (Actual); Primary Completion 2021-01-02 (Actual); Study Completion 2021-01-02 (Actual)

PRIMARY OUTCOMES:
Time required to achieve haemostasis. | 10 minutes
Number of subjects in whom haemostasis was achieved within 3 minutes after administration. | 3 minutes
Number of subjects who required surgical revision within 12 hours after the procedure for recurrent bleeding. | 12 hours

SECONDARY OUTCOMES:
Number of subjects in whom haemostasis was achieved within 2 minutes after administration. | 2 minutes
Degree of bleeding from target bleeding site | 10 minutes
Number of subjects with complications during surgery. | During a surgical procedure, an average of 1 hour
Occurrence of adverse events. | 1 month

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Hradec Králové, Hradec Králové, Czechia

IPD SHARING:
Plan to Share IPD: No